CLINICAL TRIAL: NCT07354230
Title: Open Randomised Controlled parallEl Groups Study of Gastroprotective Efficacy of Rebamipide in Patients With Atrial Fibrillation and Moderate-to-high Risk of Thromboembolic Events, Who Are Treated With Direct Oral Anticoagulants (REGATA)
Brief Title: Gastroprotective Efficacy of Rebamipide in Patients With Atrial Fibrillation Treated With DOACs
Acronym: REGATA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pirogov Russian National Research Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NIR-2021/12
Record Dates: First submitted 2025-06-11; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-05

CONDITIONS: Atrial Fibrillation (AF)
Keywords: Rebamipide; Pantoprasole; Atrial fibrillation; DOACs; Gastroprotection
MeSH Terms: conditions — Atrial Fibrillation | interventions — rebamipide; Pantoprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group Rebamipide (Experimental): 100 mg 3 times per day
  Interventions: Drug: Rebamipide 100mg
- Group Pantoprazole (Active Comparator): pantoprazol 40 mg Daily
  Interventions: Drug: Pantoprazole
- Group combination of Rebamipide and Pantoprazole (Experimental): Rebamipide 100 mg plus pantoprazol 40 mg
  Interventions: Drug: Rebamipide 100mg; Drug: Pantoprazole

INTERVENTIONS:
Drug: Rebamipide 100mg — Rebamipide 100 mg three times per day
  Arms: Group Rebamipide; Group combination of Rebamipide and Pantoprazole
Drug: Pantoprazole — 40 mg once daily
  Arms: Group Pantoprazole; Group combination of Rebamipide and Pantoprazole

SUMMARY:
The goal of this clinical trial is to learn if Rebamipide effective in gastroprotection in patients with atrial fibrillation who are treated with Direct Oral Anticoagulants (DOACs). Another point is to compare efficacy of Rebamipide and of its combination with Pantoprazole with efficacy of Pantoprazole only.

Participants will:

Take one of three variants of treatments for up to 24 weeks. Visits to the clinic wil take place for screening and then every 8 weeks.

DETAILED DESCRIPTION:
The study enrolls 210 patients with atrial fibrillation (AF) and a moderate or high risk of thromboembolic complications (>=1 point in men and >=2 points in women according to the CHA2DS2VASc scale), who receives direct oral anticoagulants (DOACs) or has indication to their dministration for prevention of thromboembolic complications and in the same time has indication for gastroprotection.

The study includes a screening period (to confirm selection criteria) and a treatment period (maximum 24 weeks), that consists of 4 visits:

* Visit 1 (randomization),
* Visit 2 and 3 - follow up,
* Visit 4 - end of study. Patients will be randomized to one of three treatment groups in a 1:1:1 ratio.
* Group Rebamipide, receiving standard therapy and rebamipide 300 mg per day
* Group Pantoprazole , receiving standard therapy and pantoprazole 40 mg per day
* Group Combination of Rebamipide and Pantoprazole, receiving standard therapy, rebamipide 300 mg per day and pantoprazole 40 mg per day Standard therapy in the study refers to the use of DOAC in accordance with applicable clinical guidelines.

Physical examination, blood pressure/heart rate measurement, Adverse Events (AEs) control, concomitant medications and compliance assessment will be performed every visit. An Esophagogastroduodenoscopy (EGD) with H. pylori detection, Lanza score assessment, GOS questionnaire, and laboratory tests (blood and stool tests) will be performed on screening and visit 4.

ELIGIBILITY:
Inclusion Criteria:

* Men and women from 18 till 80 years old
* Patients with atrial fibrillation (AF) and a moderate or high risk of thromboembolic complications (>=1 point in men and >=2 points in women according to the CHA2DS2VASc scale), receiving DOAC (rivaroxaban, apixaban or dabigatran) for the prevention of thromboembolic complications
* The following indications for the use of rebamipide and/or pantoprazole:

  * Chronic gastritis with high acidity in combination with gastroesophageal reflux disease
  * Peptic ulcer if negative test for H. pylori
  * Сhronic erosive gastritis
  * Need for

Exclusion Criteria:

* Refusal to participate in the study
* Participation in any other clinical trial or taking study drugs within 3 months before enrollment;
* Contraindications to study procedures
* Participation in the study is unsafe according to the investigator opinion.
* Admission of prohibited medication
* Pregnancy and lactation, as well as the inability to use reliable contraception in women of childbearing age
* Peptic ulcer in the acute stage
* Acute erosion on screening visit

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2022-01-11 (Actual); Primary Completion 2024-09-20 (Actual); Study Completion 2024-09-20 (Actual)

PRIMARY OUTCOMES:
Composite endpoint | up to 24 weeks
  Composite endpoint including the occurrence of any of the following events:
  * gastrointestinal bleeding;
  * symptomatic gastric or duodenal ulcer or at least 5 gastroduodenal erosions;
  * obstruction of the upper gastrointestinal tract;
  * perforation of the upper gastrointestinal tract;
  * severe dyspepsia (6-7 points according to the GOS questionnaire)

CONTACTS AND LOCATIONS:
Overall Officials: Olga Tkacheva, Principal Investigator — Pirogov Russian National Research Medical University
Locations (1):
- Russian Research and Clinical Center for Gerontology, Moscow, Russia